CLINICAL TRIAL: NCT00338897
Title: A Multicenter, Randomized, Double-Blind, Double Dummy, Parallel Group, Dose Ranging Study of Subcutaneous SR123781A With an Enoxaparin Calibrator Arm in the Prevention of Venous Thromboembolism in Patients Undergoing Elective Total Hip Replacement Surgery
Brief Title: Dose Ranging Study in Elective Total Hip Replacement Surgery
Acronym: DRIVE
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: ICD Study Director, sanofi-aventis
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: DRI5664; EudraCT : 2006-000152-41
Record Dates: First submitted 2006-06-19; First posted 2006-06-20 (Estimated); Last update posted 2008-12-10 (Estimated); Status verified 2008-12

CONDITIONS: Venous Thromboembolism
Keywords: Venous Thromboembolism; Prevention; Arthroplasty; Replacement; Hip; orthopedic surgery
MeSH Terms: conditions — Venous Thromboembolism | interventions — SR 123781A

STUDY DESIGN:
Who Masked: Participant, Investigator

INTERVENTIONS:
Drug: SR123781A

SUMMARY:
The primary objective is to:

* demonstrate the efficacy of SR123781A in the prevention of venous thromboembolism (VTE) by the demonstration of a dose-response in patients undergoing total hip replacement surgery.

The secondary objectives are to:

* evaluate the safety of SR123781A in the prevention of VTE after elective total hip replacement surgery; and
* to assess the SR123781A pharmacokinetic profile in patients undergoing elective total hip replacement surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled to undergo elective total hip replacement surgery or a revision of at least one component of a total hip replacement performed > 6 months prior to study entry

Exclusion Criteria:

* Pregnant or nursing women, or women of childbearing potential who are not using an effective contraceptive method and who do not have a negative pregnancy test performed immediately before randomization
* Known progressive malignant disease
* Ischemic stroke in the last 3 months
* Myocardial infarction (MI) in the last 3 months
* Any major orthopedic surgery in the 3 months prior to study start
* Clinical signs or symptoms of DVT or PE within the last 12 months or symptoms of post phlebitic syndrome (these conditions may confound DVT/PE assessments)
* Treatment with other antithrombotic agents within 7 days prior to surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1090 (Actual)
Dates: Start 2006-05; Primary Completion 2007-05 (Actual); Study Completion 2007-05 (Actual)

PRIMARY OUTCOMES:
The primary efficacy endpoint is a composite of total venous thromboembolic events (VTE) including VTE related deaths during the treatment period.

SECONDARY OUTCOMES:
Secondary efficacy endpoints will include all deep vein thrombosis events [DVTs] (proximal or distal) and all symptomatic VTEs (pulmonary embolisms [PEs] or DVTs)
The main safety criterion is the incidence of major bleedings occurring from the first study drug administration to 3 calendar days after the last study drug administration.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Rud Lassen, MD, Study Chair — Hoersholm Hospital, Spine Clinic, Usserod Kongevej 102, DK-2970 Hoerholm, Denmark
Locations (14):
- Sanofi-Aventis, San Isidro, Buenos Aires, Argentina
- Sanofi-Aventis, Sofia, Bulgaria
- Sanofi-Aventis, Providencia, Santiago Metropolitan, Chile
- Sanofi-Aventis, Bogotá, Colombia
- Sanofi-Aventis, Prague, Czechia
- Sanofi-Aventis, Denmark, Denmark
- Sanofi-Aventis, Helsinki, Finland
- Sanofi-Aventis, México, Mexico
- Sanofi-Aventis, Oslo, Norway
- Sanofi-Aventis, Warsaw, Poland
- Sanofi-Aventis, Bucharest, Romania
- Sanofi-Aventis, Moscow, Russia
- Sanofi-Aventis, Bromma, Sweden
- Sanofi-Aventis, Istanbul, Turkey (Türkiye)

REFERENCES:
- [Derived] Lassen MR, Dahl O, Mismetti P, Zielske D, Turpie AG. SR123781A: a new once-daily synthetic oligosaccharide anticoagulant for thromboprophylaxis after total hip replacement surgery: the DRIVE (Dose Ranging Study in Elective Total Hip Replacement Surgery) study. J Am Coll Cardiol. 2008 Apr 15;51(15):1498-504. doi: 10.1016/j.jacc.2008.03.007. PMID 18402906
- See also: Related Info — http://www.sanofi-aventis.com